CLINICAL TRIAL: NCT05847270
Title: A Randomized Controlled Study for Surgical Treatment of Irreducible Atlantoaxial Dislocation
Brief Title: Surgical Treatment of Irreducible Atlantoaxial Dislocation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Tianjin People's Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Wang Shenglin, Clinical Professor, Peking University Third Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: M2023203
Record Dates: First submitted 2023-04-14; First posted 2023-05-06 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Irreducible Atlantoaxial Dislocation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior and posterior treatment strategy (Experimental): Anterior transoral release and reduction + posterior internal fixation and bone graft fusion
  Interventions: Procedure: Anterior and posterior treatment strategy
- Simple Posterior Approach Treatment Strategy (Experimental): posterior reduction and internal fixation
  Interventions: Procedure: Simple posterior approach treatment strategy

INTERVENTIONS:
Procedure: Anterior and posterior treatment strategy — Before surgery, a large weight traction of 1/6 body weight was used to determine the reversibility of atlantoaxial dislocation. After determining that it is difficult to restore the dislocation, a technique of anterior oral release and posterior fixation fusion was used for reduction, with sequential release of the longus colli and longus capitis, the anterior longitudinal ligament, the blitateral lateral mass joints, the contracted soft-tissue mass between the odotiod and the anterior C1 tubercle, and the peri-odontoid ligaments (i.e., the alar ligaments and the apical ligament), followed by posterior internal fixation and bone grafting was used between C1 and C2 lamina.
  Arms: Anterior and posterior treatment strategy
Procedure: Simple posterior approach treatment strategy — Preceding the surgical procedure, an assessment was conducted utilizing 1/6 weight traction to ascertain the reducibility of atlantoaxial dislocation. Upon confirmation of IAAD, the chosen approach involved the utilization of a specially designed spreader, tailored to the patient's atlanto-axial joint morphology. Upon entering the joint space, the spreaders were skillfully maneuvered to gently open the joint through rotational and prying actions. Subsequently, two cages, pre-filled with autogenous bone grafts, and designed with the appropriate angle and height, were meticulously placed between the Atlanto-axial joints via a posterior approach. This procedure facilitated direct distraction and reduction of the dislocated joint. In the final step of the surgical process, stabilization was achieved by securing the atlas and axis with screws and rods. This surgical approach was selected to address the unique challenges posed by IAAD, with the aim of achieving optimal patient outcomes.
  Arms: Simple Posterior Approach Treatment Strategy

SUMMARY:
At present, there is a lack of standardized, large-scale, and high-level evidence-based medicine research on the safety and effectiveness of treatment of irreducible atlantoaxial dislocation (IAAD).Based on this, the goal of this prospective randomized controlled study is to systematically investigate the optimal surgical approach (simple posterior approach and the combined anterior and posterior approach) for managing IAAD, providing insights into the most efficacious and safest course of action. And long-term follow-up will be conducted on patients to evaluate the safety and effectiveness of different surgical methods, and to develop diagnostic and treatment standards for irreducible atlantoaxial dislocation.

DETAILED DESCRIPTION:
The choice of surgical strategies for treating irreducible atlantoaxial dislocation (IAAD) is still a controversial topic. Surgical approaches under consideration of IAAD encompass the simple posterior approach and the combined anterior and posterior approach. The former offers procedural simplicity but has inherent limitations in the extent of reduction. In contrast, the latter approach holds the potential for a more comprehensive and reliable release and reduction. However, it also presents an elevated risk of infection and surgical complexity. The choice between these two strategies remains a controversy. Based on this, the goal of this prospective randomized controlled study is to systematically investigate the optimal surgical approach for managing IAAD, providing insights into the most efficacious and safest course of action.

Six high-level centers for the treatment of IAAD participated in this randomized controlled study. After rigorous sample size analysis, we plan to recruit 260 IAAD patients into two distinct trial groups: the "Simple Posterior Surgery Group" and the "Combined Anterior and Posterior Surgery Group". By analysing the comprehensive radiological assessment, the systematic tracking of neurological function improvement, meticulous evaluation of specific adverse events and a 12 month post-surgery follow-up we will systematically investigate the optimal surgical approach for managing IAAD.

Besides, this research endeavor has received full ethical clearance from the Peking University Third Hospital (PUTH) Medical Science Research Ethics Committee (IRB00006761-M2023203). All enrolled participants will provide informed consent voluntarily.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants encompass individuals within the age range of 0 to 80 years, without regard to gender.
2. Patients who have received a diagnosis of irreducible atlantoaxial dislocation (IAAD) based on preoperative imaging and skull traction evaluation, with a traction weight equivalent to 1/6 of their body weight following anesthesia. These patients are candidates for surgical intervention.
3. Participants who have provided informed consent either in person or through their legal representative (the principal).

Exclusion Criteria:

1. Individuals with concomitant medical conditions or diseases that significantly impact surgical treatment, such as malignant metastasis or infectious diseases, will be excluded from the study.
2. Critically ill patients, who are not suitable candidates for surgical intervention, will also be excluded.
3. Patients who actively decline to participate in this research project will not be included in the study cohort.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Decompression Rate | 12 months
  Effective spinal cord decompression on MRI, and the arachnoid space between the spinal cord and the odontoid process can reappear.
Bone Graft Fusion Rate | 12 months
  Evaluation of the proportion of patients exhibiting successful bone fusion between the atlas and axis will be conducted through postoperative three-dimensional CT examinations of the cervical spine. The bone graft fusion rate will be determined by calculating the number of patients with evident fusion relative to the total number of patients enrolled.
Atlantoaxial Reduction Rate | 12 months
  To gauge the effectiveness of the surgical interventions in achieving atlantoaxial reduction, postoperative CT scans of the head and neck will be conducted. Measurements will be taken of the distance between the odontoid process and key reference lines, including Chamberlain's line (CL), Wackenheim line (WL), McRae line (ML), and atlantodental interval (ADI). The reduction rate will be calculated by comparing the postoperative measurements to the preoperative values, expressed as a ratio.

SECONDARY OUTCOMES:
Incidence of Adverse Events (12 Months After Surgery) | 12 months
  The primary focus of evaluation is on the incidence of adverse events occurring within the 12-month post-surgery period. This metric is defined as the proportion of adverse events that manifest during the study's duration relative to the total number of patients enrolled. Adverse events encompass a range of critical factors, including but not limited to: Neurological deterioration, Incision infection, Vascular injury, Airway obstruction, Poor reduction, Unplanned readmission and re-surgery, Internal fixation failure, Fusion failure, Surgical-related lower cervical spine deformities.
Improvement Rate of Quality of Life (12 Months After Surgery) | 12 months
  The quality of life for each patient will be assessed using the SF-12 Health Survey. The improvement rate in quality of life will be calculated based on the preoperative and postoperative differences in SF-12 scores. This indicator offers insights into the impact of surgical interventions on patients' overall well-being and quality of life, providing a vital perspective on treatment effectiveness.
Improvement of Neurological Function | 12 months
  To assess the extent of neurological function improvement, patients' JOA scores one year after surgery will be compared with their preoperative scores. The JOA improvement rate will be calculated based on the cervical JOA score, employing the Hirabayashi method formula: JOA Improvement Rate = (Postoperative JOA Score - Preoperative JOA Score) / (17 - Preoperative JOA Score) * 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No